CLINICAL TRIAL: NCT05736952
Title: Oral Topotecan Combined With Anlotinib in Patients With Platinum-resistant Recurrent Ovarian Cancer：
Brief Title: Oral Topotecan Combined With Anlotinib in Patients With Platinum-resistant Recurrent Ovarian Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Program changed
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XH-22-015
Record Dates: First submitted 2023-02-12; First posted 2023-02-21 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-02

CONDITIONS: Platinum-resistant Ovarian Cancer
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral Topotecan Combined With Anlotinib (Experimental)
  Interventions: Drug: Oral Topotecan Combined With Anlotinib

INTERVENTIONS:
Drug: Oral Topotecan Combined With Anlotinib — Topotecan hydrochloride capsules: 2 mg, once daily, oral with dinner for 5 days, discontinued for 16 days, that is, 21 days (3 weeks) as a course of treatment, a total of 6 courses of administration.；Anlotinib hydrochloride capsules: 10mg once a day, oral before breakfast, continuous administration for 14 days, discontinuation for 7 days, that is, 21 days (3 weeks) as a course of treatment.

SUMMARY:
The goal of this clinical trial is to evaluate the treatment of topotecan hydrochloride capsules combined with anlotinib hydrochloride capsules in Patients with platinum-resistant recurrent epithelial ovarian cancer. The main questions it aims to answer are: to assess the objective response rate (ORR), progression-free survival (PFS), disease control rate (DCR), duration of response (DOR), overall survival (OS) and safety of topotecan hydrochloride capsules combined with anlotinib hydrochloride capsules in patients with platinum-resistant recurrent epithelial ovarian cancer.The treatment of participants： Topotecan hydrochloride capsules: 2 mg, once daily, oral with dinner for 5 days, discontinued for 16 days, that is, 21 days (3 weeks) as a course of treatment, a total of 6 courses of administration.；Anlotinib hydrochloride capsules: 10mg once a day, oral before breakfast, continuous administration for 14 days, discontinuation for 7 days, that is, 21 days (3 weeks) as a course of treatment. Receiving optimal supportive care at the same time until disease progression/death/intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 18 years old;
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
3. The pathological type is epithelial ovarian cancer: high-grade serous, clear cell, endometrium-like; or fallopian tube cancer, primary peritoneal cancer;
4. After surgery, the patient received ≥ 2 lines of chemotherapy,Platinum resistant ovarian cancer (defined as relapsing within 6 months after the last administration of platinum-based chemotherapy);
5. Clinical recurrence with measurable lesions (with imaging evidence);
6. Estimated survival≥ 3 months;
7. The main organs function well, and the examination indicators meet the following requirements: 1) Routine blood test: hemoglobin ≥ 90 g/L (no transfusion within 14 days); Neutrophil count≥ 1.5×109/L; Platelet count≥ 80×109/L; 2) Biochemical examination: Total bilirubin ≤1.5×ULN (upper limit of normal); Blood valley alanine aminotransferase (ALT) or blood valley aminotransferase (AST) ≤ 2.5×ULN; ALT or AST ≤ 5×ULN if liver metastases are present; Serum creatinine ≤ 1.5×ULN or endogenous creatinine clearance ≥ 50 ml/min (Cockcroft-Gault formula);
8. Good compliance, family members agree to cooperate with survival follow-up.

Exclusion Criteria:

1. Have other malignant tumors at the same time, except for malignant tumors that have been cured or stabilized;
2. Pregnant or lactating women;
3. Participated in clinical trials of other drugs within six months;
4. Have a variety of factors that affect oral drugs (such as inability to swallow, chronic diarrhea and intestinal obstruction, etc.);
5. Any bleeding event with a severe grade of 3 or above in CTCAE 4.0 within 4 weeks prior to screening;
6. Patients with known central nervous system metastases or history of central nervous system metastases before screening;
7. Patients with hypertension who cannot be well controlled by single antihypertensive drugs (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg); Patients with a history of unstable angina; Patients with a new diagnosis of angina within 3 months before screening or a myocardial infarction event within 6 months before screening; Arrhythmias require long-term use of antiarrhythmic drugs and New York Heart Association grade ≥ II cardiac insufficiency;
8. Long-term unhealed wounds or incompletely healed fractures;
9. Previous organ transplantation history;
10. Imaging shows that the tumor has invaded important blood vessels or the investigator judges that the patient's tumor has a high possibility of invading important blood vessels during treatment and causing fatal hemorrhage;
11. Coagulation dysfunction (prothrombin time>16s, Activated partial thromboplastin>43s, thrombin time>21s, fibrinogen<2g/L), with bleeding tendency (14 days before randomization must meet: INR within normal value without anticoagulant); Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogues; Under the premise of the international normalized ratio (INR) of prothrombin time (INR) ≤ 1.5, the use of low-dose warfarin (1 mg orally once daily) or low-dose aspirin (not exceeding 100 mg daily) for prophylactic purposes is permitted;
12. Screen for arteriovenous thrombotic events within one year before, such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis (except for venous thrombosis caused by venous catheterization with chemotherapy in the early stage of chemotherapy and judged to have been cured by the investigator) and pulmonary embolism;
13. Those who have a history of psychotropic substance abuse and cannot quit or have mental disorders;
14. Have a history of immunodeficiency, or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;
15. According to the judgment of the investigator, there are serious concomitant diseases that endanger the safety of patients or affect the completion of the study;
16. History of surgical procedures within 28 days;
17. History of abdominal fistula or gastrointestinal perforation within 28 days;
18. Those who may receive other systemic anti-tumor therapy or plan to undergo ovarian cancer debulking surgery during the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | one year

SECONDARY OUTCOMES:
progression-free survival (PFS) | one year
disease control rate (DCR) | one year
duration of response (DOR) | one year
overall survival (OS) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Xipeng Wang, Dr, Study Director — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided